CLINICAL TRIAL: NCT01790165
Title: A Phase II Open Label Multiple-Dose Study of the Safety and Pharmacokinetics of TDT 067 Under Conditions of Maximal Use in Subjects With Distal Subungual Onychomycosis of the Toenails
Brief Title: TDT 067 Open Label Multi-Dose Onychomycosis Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celtic Pharma Development Services (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: CL-067-II-02
Record Dates: First submitted 2010-03-18; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Open Label; PK
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDT067 (Experimental): Active treatment
  Interventions: Drug: TDT067 and Lamisil
- Placebo (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: TDT067 and Lamisil — Topical administration of TDT067 and single oral administration of 250 mg Lamisil tablet
  Other Names: Lamisil
  Arms: TDT067

SUMMARY:
The aim of this study is to establish a clinical bridge to Lamisil® tablets by conducting a clinical pharmacokinetic (PK) study comparing the systemic exposure of a Lamisil® tablet with that of with TDT 067 under maximal use conditions.

Under maximal use conditions in onychomycotic subjects, the aim is to confirm that there are significantly lower plasma levels of terbinafine and its major metabolites after a topical administration of TDT 067 for 28 days in comparison with a single oral 250 mg Lamisil® tablet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18 and 65 years of age inclusive, of any race, and of either sex.
* Male subjects only: Male subjects must use a reliable form of contraception during their participation in the trial and for 3 months after their last dose of study drug.
* Female subjects only: Either of non-childbearing potential (i.e. either surgically sterilized or post menopausal) or must be using adequate contraception, have a negative pregnancy test prior to start of dosing, and must agree to continue to use this method of contraception until 3 months after the last dose. Acceptable contraceptive methods are oral contraceptive, IUD, or diaphragm with spermicide (unless anatomically sterile).
* Subjects must be in good general health as confirmed by a medical history and physical examination.
* Subjects must have 2 big toes with nails that have the potential to be clipped to provide nail samples.
* Subjects must have clinically diagnosed distal subungual onychomycosis of the toenails; at least 5 nails in total must present with onychomycotic signs (onycholysis, subungual hyperkeratosis) including extensive involvement (≥50%) of both large nails and mycological confirmation (positive KOH microscopy) from 1 of the large nails.
* Subject must sign a statement of informed consent.
* Subjects must be able to understand the requirements of the study, abide by the restriction, and return for all of the required examinations

Exclusion Criteria:

* Subjects lacking any toes.
* Subjects with known hypersensitivity to terbinafine or any of the excipients in the TDT 067.
* Subjects with symptomatic tinea pedis requiring treatment.
* Subjects with any medical, neurological, or psychiatric conditions that in the opinion of the Investigator would make the subject unsuitable for enrollment onto the study.
* Subjects with chronic or active liver disease, as well as subjects with elevated liver function tests above normal for the testing laboratory.
* Subjects with renal impairment (creatinine clearance ≤50 mL/min).
* Subjects who have received terbinafine tablets within 12 months or topical terbinafine (cream, solution/spray, or gel) within 6 months prior to screening visit; subjects who have received other oral antifungals within 4 months or other topical antifungals within 1 month.
* Subjects who have participated within the previous 3 months in a clinical trial for the systemic or topical treatment of onychomycosis.
* Subjects being treated with rifampin or cimetidine.
* Subjects being treated with an investigational drug within 1 month prior to study start.
* Subjects with psoriasis or history of psoriasis.
* Subjects with nail dystrophy or other nail abnormalities other than onychomycosis.
* Subjects with serious concurrent disease that might prevent completion of the trial.
* Subjects who are pregnant (confirmed by pregnancy test) or who plan to become pregnant within the study timeframe or who are nursing.
* Subjects who cannot read, understand, or sign the informed consent form or the instructions for applying and removing the study formulations.
* Subjects who cannot apply the product to their toenails.
* Subjects who do not wish to provide nail clippings.
* Subjects who cannot or will not provide adequate blood and urine samples.
* Subjects using any nail polish products or other nail cosmetic products on any of the toenails designated for treatment within 7 days prior to the start of treatment and who are unwilling to discontinue use of these products for the duration of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PK | 35 days
  Cmax, Tmax, AUC0-12, AUC0-24, Cmax Ratio (day 28/day 35) were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tschen, MD, Principal Investigator — Academic Dermatology Assoc